CLINICAL TRIAL: NCT06686706
Title: Comparing the Effectiveness of Instrumental Assisted Soft Tissue Mobilization (IASTM) and Kinesio Taping on Foot Functional Status and Quality of Life (QOL) in Plantar Fasciitis
Brief Title: Effects of IASTM and Kinesiotaping in Plantar Fascitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Riphah/RCRAHS/REC/MS-PT/01943
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Plantar Fascitis
Keywords: Plantar Fascitis; IASTM; Graston technique; Kinesio Taping

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IASTM Group (Experimental): Instrumental Assisted Soft Tissue Mobilization
  Interventions: Other: IASTM
- KT Group (Experimental): Kinesiotaping
  Interventions: Other: KT group

INTERVENTIONS:
Other: IASTM — Graston therapy-8 min per session
  Procedure:
  The patient will be lying down with their knee bent 30 degrees. After a 5-minute ultrasound treatment and static stretching exercises.Treatment will be administered using the Graston tool (using the sweep approach). Applying a moderate amount of effort from the medial side of the heel to the metatarsals and from the metatarsals to the medial side of the heel, to-and-fro stroking at a 60° angle will be done on the sole of the foot for approximately eight minutes (60-70 strokes per minute with a 5- to 10-second rest interval. A cold pack will be used for five minutes after therapy. The GT session will last approximately 30 minutes.
  Conventional Therapy:
  Therapeutic ultrasound for 5 min Stretching of plantar fascia 5 reps with 10 sec hold) Cold therapy for 5 min Functional status and Quality of Life (QOL) will be assessed before and after treatment of 4 weeks using using tools.
  Intervention will be conducted once a week for 4 weeks.
  Arms: IASTM Group
Other: KT group — Kinesio tapping (left there for 3 days)
  Procedure:
  We will use a standard 2" (5 cm) kinesiology tape. Fascia tape will be applied to the plantar fascia, and it will be left there for three days. For four weeks, it will be applied once a week. The patient will be in a prone position, lying with the ankle joints in a neutral position while applying tape. With the toes extended against the bed or ground. The tape will be marked on the Achilles tendon. It will be cut longitudinally into five slices of equal width. It will be applied to the forefoot by stretching it by 25%. The last strap will be applied with gentle compression across the bases of the five slices beneath the foot and wrapped around the rear foot.(5) Conventional Therapy Therapeutic ultrasound for 5 min Stretching of plantar fascia 5 reps with 10 sec hold) Cold therapy for 5 min
  Arms: KT Group

SUMMARY:
The Objective of the study is to compare the effectiveness of Instrumental Assisted Soft Tissue Mobilization (IASTM) and Kinesio taping for improving foot functional status and Quality of Life (QOL) in patients with Plantar Fasciitis. The study will be randomized controlled Trial including 2 experimental groups and 19 participants in each group

DETAILED DESCRIPTION:
Plantar fasciitis is one of the most frequent foot problems that affects 11 to 15% of people with foot problems between the ages of 25 and 65 years old who walk and stand for a long time at the workplace. It is a chronic inflammatory disorder that occurs at the medial calcaneal tuberosity as a reaction to repeated injury or exposure to tremendous pressures at the calcaneus insertion, causing inflammation and plantar fascia tears. It is one of the most common causes of heel pain that affects more than 3 million people in the United States alone every year. It is thought to affect 4-10% of the general population.

The thick band of connective tissue that runs the length of the foot and supports the arch is called the plantar fascia. It plays a vital role in maintaining arch of foot and absorbing shock while weight bearing activities. It has three components: a thinner medial and lateral component, and a thicker central component. The plantar fascia forms the longitudinal arch of the foot by inserting into each metatarsal head after emerging from the posteromedial calcaneal tuberosity. Some reported cases of plantar fasciitis are the result of biomechanical failure that provides tension along the plantar fascia.

Risk factors that cause damage to the plantar fascia include excessive foot pronation, jogging, obesity, prolonged standing, and inadequate ankle dorsiflexion. Limited ankle dorsiflexion, a body mass index higher than 27 kg per m2 and spending the most of the workday on one's feet are risk factors for developing plantar fasciitis in non-athletes. The most common symptom is painful medial plantar heel pain in the first few steps after sitting or sleeping. The pain usually goes away after further ambulation, but it can return with continued weightbearing.

Traditionally, it was believed that plantar fasciitis is induced by mechanical damage in which the plantar fascia was subjected to excessive tensile strain, which caused tiny tears and persistent inflammation. According to current theories, plantar fasciitis develops through a deterioration of fascia, which is why it is sometimes referred to as Fasciosis rather than Fasciitis, where maximum stress is the main factor in the etiology. Gap junctions between fibrocytes specifically perceive the increased fascial stress, which subsequently mediates alterations in the extracellular matrix, leading to myxoid deterioration and breakage of the plantar fascia.

Among the conservative therapy approaches for Plantar Fasciitis (PF) include activity modification, ice massage, stretching exercises, orthotics, oral analgesics, and corticosteroid injections. Low-level laser therapy, ultrasound therapy, and extracorporeal shockwave therapy (ESWT) are further treatment options for chronic plantar fasciitis (LLLT). Clinicians commonly employ a form of manual treatment called soft tissue mobilization/manipulation (STM) to lessen the pain and dysfunction brought on by musculoskeletal disorders. 87% of doctors use manual therapy on a daily basis. Instrumental Assisted Soft Tissue Mobilization (IASTM's) myofascial restriction, which is based on James Cyriax's soft tissue mobilization, gained increased attention recently. It has been proposed that IASTM acts as a neuromodulatory factor in pain regulation by activating mechanosensitive neurons found in the soft tissues that have been treated. The deformation of the skin may result in a reduction in the activity of fiber neurons, potentially producing an analgesic effect.

KT is an elastic therapeutic taping tool consisting of mainly of cotton, introduced by Dr. Kenso Kase in 1970s. It is lightweight, waterproof, breathable, and available in wide range of colors, types, lengths, textures. These features allow for multiple day wear and a constant pulling force on the skin. This pulling force to the skin on which kinesiotape is applied is thought to improve blood and lymphatic circulation, resulting in pain and edema relief. Following assessments and instructions from healthcare professionals, KT can be directly fixed to target tissue with combination of cuts (e.g. Y, I, X tape), tensions (% of stretch) and directions (e.g. muscle insertion to origin). Wearing KT maintain effect for 3-5 days, ideally following the 24 hours application rule based on skin condition. KT's therapeutic effects include increasing subcutaneous space, stimulating skin sensory receptors, supporting mechanical behavior, promoting micro circulation, and relieving pain in musculoskeletal disorders, improving proprioception stability, range of motion, and quality of life.

Previous studies have primarily focused on the effectiveness of Kinesio tapping solely on pain, function and quality of life in plantar fasciitis. In the past study, it was suggested to use conventional therapy along with Kinesio tape. Conventional therapies aim to alleviate pain, reduce inflammation and restore normal function. Thus, investigating the effectiveness of combining conventional therapy with Kinesio tapping in improving foot function and QOL in patients with plantar fasciitis. This research aims to fill the existing gap in literature by providing evidence-based guidance on optimal management approach for plantar fasciitis.This study will contribute in describing that which technique is best in management of plantar fasciitis and define the effects of both techniques on improving functional status and QOL.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Age Range of 20-40 years
* Standing > 8 hours a day
* Positive Windlass test
* Patients who experience pain on medial tuberosity of the calcaneus on palpation.
* Pain during the initial steps that lessened after a few steps but aggravated by increased activity

Exclusion Criteria:

* History of ankle or foot surgery
* Patients with inflammatory conditions like cancer, rheumatoid arthritis, ankle and foot bursitis.
* Foot related complications after fracture
* Patients receiving corticosteroid injections

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-12-13 (Estimated); Study Completion 2024-12-13 (Estimated)

PRIMARY OUTCOMES:
Foot and Ankle Outcome Score (FAOS): | 4 weeks
  FAOS is a 42-item questionnaire divided into 5 subscales pain (9 items), other symptoms (7 items), ADL (17 items), sport/recreation (5 items) and quality of life (4 items). A five-point Likert scale, with 0 denoting no problem, 1 mild, 2 moderate, 3 severe, and 4 extreme problems, is used to grade each item. Each subscale's total score is summed together and divided by the subscale's maximum score, to determine the score for each subscale. A scale of 0 to 100 is created from the normalized score, where 100 represents no problems and 0 represents severe problems.
SF-12 | 4 weeks
  A short health survey-12 version 2 is used to measure quality of life (SF-12 V.2). The patients' overall health and quality of life will be assessed using this questionnaire. There are twelve questions on the assessment form, and the answers can be used to score eight different areas of health. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning. A score of 50 or less on the PCS-12 has been recommended as a cut-off to determine a physical condition; while a score of 42 or less on the MCS-12 may be indicative of 'clinical depression'. There are two categories on the SF-12 V.2 surveys: Mental and Physical health. Cronbach's alpha values, which ranged from 0.60 to 0.87, supported the dependability and internal consistency.

CONTACTS AND LOCATIONS:
Overall Officials: Shumaila Parveen, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Bahria Active, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang J, Nie D, Rocha JL, Hogan MV, Wang JH. Characterization of the structure, cells, and cellular mechanobiological response of human plantar fascia. J Tissue Eng. 2018 Oct 3;9:2041731418801103. doi: 10.1177/2041731418801103. eCollection 2018 Jan-Dec. PMID 30302189